CLINICAL TRIAL: NCT00852527
Title: Evaluation of VA's TBI Clinical Reminder And Secondary Level Evaluation
Brief Title: Evaluation of VA's Traumatic Brain Injury (TBI) Clinical Reminder and Comprehensive TBI Evaluation (CTBIE)
Acronym: TBI
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: SDR 08-377
Record Dates: First submitted 2009-02-25; First posted 2009-02-27 (Estimated); Results first posted 2014-12-05 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-08

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Screening; Diagnosis; Rehabilitation Outcome
MeSH Terms: conditions — Brain Injuries, Traumatic; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects with mild TBI: Presence of mild TBI defined by positive reference test
- Subjects without mild TBI: Absence of mild TBI defined by negative reference test

SUMMARY:
The purpose of the proposed study is to determine the clinical validity and reliability of the VA's Traumatic Brain Injury (TBI) Clinical Reminder Screen and the Comprehensive TBI Evaluation used to screen for mild traumatic brain injury. Examining the reliability of the two screens will determine whether they are dependable. Verifying the clinical validity is important because valid screening and evaluation of mild TBI leads to accurate diagnosis and timely treatment. Accurate screening also improves clinical efficiency and ensures that resources are provided to those who need them most. The project findings are expected to advance the science of screening and diagnosis of a mild TBI event.

DETAILED DESCRIPTION:
A. Anticipated Impacts on Veterans' Healthcare: Determining the clinical validity of the VA's TBI Clinical Reminder Screen and Comprehensive TBI Evaluation is critical because valid screening and evaluation of mild traumatic brain injury (mTBI) leads to accurate diagnosis and timely treatment. Accurate screening improves clinical efficiency and ensures that resources are provided to those who need them most. The project findings are expected to advance the science of screening and diagnosis by clarifying whether symptoms are consistent with post-concussion syndrome due to an mTBI event. Findings are also expected to inform the development of the next generation of VA screening instruments for mild TBI.

B. Project Background/Rationale: Traumatic brain injury (TBI) is a leading injury among military personnel serving in the Operation Enduring Freedom/ Operation Iraqi Freedom (OEF/OIF) combat theaters due largely to improvised explosive devices. While TBI severity ranges from mild to severe, mTBI is particularly difficult to identify, diagnose and treat. The VA modified a version of the Defense and Veterans Brain Injury Center (DVBIC) tool, which is used to screen returning OEF/OIF service members. The VA's modified screen, the TBI Clinical Reminder Screen, is used to screen a slightly different population. Therefore, results of the validity study for the DVBIC tool are not directly applicable. As a result, the General Accountability Office (GAO) recommended the VA expeditiously evaluate the clinical validity and reliability of its TBI screening tool.

C. Primary Study Objectives are: (1) Develop the Diagnostic Assessment Battery for use as a proxy gold standard, and (2) Evaluate and compare the performance characteristics of the TBI Clinical Reminder Screen and the Comprehensive TBI Evaluation using the Diagnostic Assessment Battery. These objectives will be realized via: (a) An examination the performance characteristics (diagnostic validity) of the TBI Clinical Reminder Screen and the Comprehensive TBI Evaluation relative to the Diagnostic Assessment Battery to determine sensitivity and specificity, (b) Determining whether false positives and/or false negatives are related to Post Traumatic Stress Disorder (PTSD) and how the performance characteristics of the tests differ for PTSD, (c) Ascertaining the concordance among measures of functional impairment, the TBI Clinical Reminder Screen and the Comprehensive TBI Evaluation, (d) Establishing the concurrent validity between the diagnosis of presence or absence of post-concussion syndrome due to mTBI and measures of functional impairment, (e) Verifying the test/retest reliability for the TBI Clinical Reminder Screen and the Comprehensive TBI Evaluation and (f) Identifying whether clusters of symptoms or subjects reporting similar patterns of symptoms correspond with clinical sub-groups (e.g., mTBI with PTSD, PTSD alone).

D. Project Methods: An online Delphi process and will be conducted with mTBI experts to inform the development of the Diagnostic Assessment Battery. A sample of 500 OEF/OIF veterans will be recruited over 12-months at three VA Polytrauma Network Sites. The OEF/OIF veterans will have symptoms consistent with either a mild TBI event (True Positive) or symptoms inconsistent with such an event (True Negative). All subjects will be assessed by research clinicians using the TBI Clinical Reminder Screen, the Comprehensive TBI Evaluation and the Diagnostic Assessment Battery. Analysis will determine the sensitivity and specificity as well as the test/retest reliability of the TBI Clinical Reminder and the Comprehensive TBI Evaluation. The performance characteristics for the Diagnostic Assessment Battery will be ascertained and used to further our understanding of how best to distinguish mTBI symptoms from related and/or comorbid conditions (e.g., PTSD, anxiety, and depression).

ELIGIBILITY:
Inclusion Criteria:

Patients included are those service members or Veterans who have been deployed in the OEF/OIF conflict and have screened positive or negative on the TBI Clinical Reminder.

Exclusion Criteria:

Exclusion criteria include those service members or Veterans diagnosed with a moderate to severe TBI or a psychiatric disorder unrelated to TBI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Operation Enduring Freedom/ Operation Iraqi Freedom (OEF/OIF) Veterans
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judi L Babcock-Parziale, PhD, Principal Investigator — Southern Arizona VA Health Care System, Tucson, AZ
Locations (3):
- United States (3):
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - VA Medical Center, Lexington, Lexington, Kentucky

REFERENCES:
- [Result] Pape TL, High WM Jr, St Andre J, Evans C, Smith B, Shandera-Ochsner AL, Wingo J, Moallem I, Baldassarre M, Babcock-Parziale J. Diagnostic accuracy studies in mild traumatic brain injury: a systematic review and descriptive analysis of published evidence. PM R. 2013 Oct;5(10):856-81. doi: 10.1016/j.pmrj.2013.06.007. PMID 24160300
- [Result] Shandera-Ochsner AL, Berry DT, Harp JP, Edmundson M, Graue LO, Roach A, High WM Jr. Neuropsychological effects of self-reported deployment-related mild TBI and current PTSD in OIF/OEF veterans. Clin Neuropsychol. 2013;27(6):881-907. doi: 10.1080/13854046.2013.802017. Epub 2013 Jun 11. PMID 23755991
- [Result] Combs HL, Berry DT, Pape T, Babcock-Parziale J, Smith B, Schleenbaker R, Shandera-Ochsner A, Harp JP, High WM Jr. The Effects of Mild Traumatic Brain Injury, Post-Traumatic Stress Disorder, and Combined Mild Traumatic Brain Injury/Post-Traumatic Stress Disorder on Returning Veterans. J Neurotrauma. 2015 Jul 1;32(13):956-66. doi: 10.1089/neu.2014.3585. Epub 2015 Feb 26. PMID 25350012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 456 participants were selected from three VA Polytrauma Network Sites and represent urban, suburban, and rural catchment areas. 438 completed all assessments necessary for analysis.
Groups:
- Positive Mild TBI: Participants who screened positive on the TBI Clinical Reminder Screen
- Negative Mild TBI: Participants who screened negative on the TBI Clinical Reminder Screen
Period: Overall Study
Arm/Group | Positive Mild TBI | Negative Mild TBI
Started | 196 | 242
Completed | 196 | 242
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of participants consented and enrolled.
Groups:
- OEF/OIF Veterans: Operation Enduring Freedom /Operation Iraqi Freedom (OEF/OIF) Veterans seeking care at one of three VA Polytrauma Network Sites (PNS) who screen positive or negative for mild traumatic brain injury.
Arm/Group | OEF/OIF Veterans
Number analyzed (Participants) | 438
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 33 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 392
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 39
  White | 330
  Other | 14
  Multi-Racial | 30
  Unknown | 25
Region of Enrollment [Number; unit: participants] — A sample of 438 OEF/OIF Veterans enrolled across the three sites (n Tucson = 131; n Hines = 134; n Lexington = 173).
  participants
    United States | 438

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy of the TBI Clinical Reminder Screen (TCRS)
Description: Patients were initially assessed with the TBI Clinical Screen at their local VA. To assess the diagnostic accuracy of the TCRS, a dual-criterion approach was used. The VA Comprehensive TBI Evaluation (CTBIE), a secondary evaluation, served as the first criterion and the Structured TBI Diagnostic Interview (STDI) as the second criterion.
Time Frame: All OEF/OIF Veterans to receive TCRS upon enrollment in VA
Population: Although 456 participants were consented and enrolled in the study, data for 13 participants had missing assessment data and another 5 were determined to have moderate TBI resulting in 438 cases for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Veterans Assessed With the Comprehensive TBI Evaluation | Veterans Assessed With the Structured TBI Diagnostic Interview
Number analyzed (Participants) | 438 | 438
Percentage of participants
  Sensitivity | 71 [64 to 78] | 79 [73 to 84]
  Specificity | 74 [68 to 79] | 85 [80 to 90]
  Positive Predictive Value | 32 [28 to 37] | 49 [41 to 57]
  Negative Predictive Value | 94 [92 to 95] | 96 [95 to 97]

ADVERSE EVENTS:
Groups:
- OEF/OIF Veterans: No adverse events.
Arm/Group | OEF/OIF Veterans
Serious Adverse Events (participants affected / at risk) | 0/433
Other Adverse Events (participants affected / at risk) | 0/433

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes